CLINICAL TRIAL: NCT05409131
Title: Efficacy and Safety of the Omnipod 5 System Compared to Pump Therapy in the Treatment of Type 1 Diabetes: a Randomized, Parallel-group Clinical Trial
Brief Title: Omnipod 5 System Compared to Pump Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insulet Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP5-003 (G6 CSII)
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: T1D; Omnipod; Automated Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention Arm (Active Comparator): Omnipod 5 System with Dexcom G6 continuous glucose monitoring system
  Interventions: Device: Omnipod 5 System
- Control Arm (No Intervention): Participant's current insulin pump with Dexcom G6 continuous glucose monitoring system

INTERVENTIONS:
Device: Omnipod 5 System — Omnipod 5 System automates insulin delivery based on information received from the continuous glucose monitoring system every 5 minutes.
  Arms: Intervention Arm

SUMMARY:
Subject will undergo a 14-day outpatient, standard therapy phase during which sensor and insulin data will be collected. This will be followed by a 90-day outpatient phase where subjects will either use the Omnipod 5 system or continue to use their personal insulin pump with the study provided continuous glucose monitoring system.

Participants in France will be offered an optional extension of 12 months of Omnipod 5 System use.

DETAILED DESCRIPTION:
This is an outpatient study that consists of two phases, Phase 1 and Phase 2. There will be approximately 8 study visits conducted in person or via telehealth.

Phase 1 is a 14-day period to collect baseline sensor and insulin data where subjects will manage their diabetes at home per their usual routine using the study continuous glucose monitoring system.

Phase 2 is a 90-day period where subjects will be randomized into one of two groups. One group will use the Omnipod 5 system and the other group will continue to use their personal insulin pump with the study continuous glucose monitoring system.

Following the 90-day outpatient phase, participants in France will be offered the option to transition to use the CE-marked commercial Omnipod 5 System for an additional 12 months with the French interface.

ELIGIBILITY:
Inclusion Criteria:

1. Age at time of consent 18-70 years of age
2. Diagnosed with type 1 diabetes for at least 1 year. Diagnosis is based on investigator's clinical judgment.
3. On pump therapy for ≥ 3 months prior to screening and familiar with pump therapy concepts such as basal and bolus insulin delivery, and carbohydrate counting. Participants using automated insulin delivery (AID) devices, including devices with predictive low glucose suspend (PLGS), in the 3 months prior to screening, will be excluded from participating.
4. A1C 7.0-11.0% by point-of-care taken at screening visit
5. Willing to use and obtain U-100 insulin: (either insulin aspart (Novolog, NovoRapid), or insulin lispro (Humalog, Admelog)), as the primary insulin treatment
6. Must have a smartphone that supports the Dexcom app download and participants must be willing to use the app throughout the study
7. Investigator has confidence that the participant can safely operate all study devices and can adhere to the protocol
8. Willing to wear the system continuously throughout the study
9. Willing and able to sign the Informed Consent Form (ICF)

Exclusion Criteria:

1. Any medical condition, such as untreated malignancy, unstable cardiac disease, unstable or end-stage renal failure, eating disorders, or other conditions which in the opinion of the investigator, would put the participant at an unacceptable safety risk
2. History of severe hypoglycemia in the past 6 months
3. History of diabetic ketoacidosis (DKA) in the past 6 months, unrelated to an intercurrent illness or infusion set failure
4. Blood disorder or dyscrasia within 3 months prior to screening, including use of hydroxyurea, which in the investigator's opinion could interfere with determination of HbA1C.
5. Currently on systemic steroids or intends to receive systemic steroid treatment during study participation, including stable treatment for adrenal insufficiency. Inhaled, ophthalmic, topical, joint injection, and other locally applied steroids are allowed.
6. Unable to tolerate adhesive tape or has any unresolved skin condition in the area of sensor or pump placement
7. Use of non-insulin anti-hyperglycemic medication other than metformin, in the 12 weeks prior to the Baseline Visit. Participants taking metformin should remain on a steady dose during study participation.
8. Pregnant or lactating, or is a woman of childbearing potential and not on acceptable form of birth control (acceptable forms of contraception include abstinence, barrier methods such as condoms, hormonal contraceptives, intrauterine device, surgical sterilization such as tubal ligation or hysterectomy, or vasectomized partner)
9. Participation in another clinical study using an investigational drug or device within 30-days or 5 half-lives (whichever is longer) prior to screening, or intends to participate in any other study during this study period
10. Unable to follow clinical protocol for the duration of the study or is otherwise deemed unacceptable to participate in the study per the investigator's clinical judgment
11. Participant is an employee of Insulet, an Investigator or Investigator's study team, or immediate family member of any of the aforementioned

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2025-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Weinstock, MD, Study Chair — State University of New York - Upstate Medical University; Eric Renard, Pr, Study Chair — Lapeyronie Montpellier University Hospital
Locations (14):
- United States (10):
  - Stanford University School of Medicine, Palo Alto, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - University of Colorado Denver, Denver, Colorado
  - Atlanta Diabetes, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Joslin Diabetes Center, Boston, Massachusetts
  - State University of New York, Upstate Medical University, Syracuse, New York
  - Diabetes & Glandular Disease Clinic, P.A. (DGD Clinic), San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- France (4):
  - Hopital Sud-Francilien, Corbeil-Essonnes
  - Hospices Civils de Lyon - Centre du diabete Diab-eCare, Lyon
  - CHRU de Montpellier, Hopital Lapeyronie - Departement d'endocrinologie, Diabete, Nutrition, Montpellier
  - Hopital Lariboisiere - Centre Universitaire du Diabete et de ses Complications, Paris

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 132 | 62
Completed | 131 | 21
Not Completed | 1 | 41

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 132 | 62 | 194
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (14) | 36 (13) | 36 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 38 | 116
  Male | 54 | 24 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to privacy laws, race and ethnicity were reported by participants in the U.S. only.
  Two participants identified as "Other race", so their results are included in the "Unknown or Not Reported" row.
  Participants
    number analyzed (Participants) | 80 | 38 | 118
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 1 | 2 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 4 | 3 | 7
    White | 70 | 29 | 99
    More than one race | 2 | 2 | 4
    Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 80 | 38 | 118
  France | 52 | 24 | 76
BMI (kg/m^2) [Mean (Standard Deviation); unit: (kg/m^2)] | 26.6 (4.8) | 25.4 (4.1) | 26.2 (4.6)
HbA1c at Screening [Mean (Standard Deviation); unit: Percentage] | 8.5 (0.8) | 8.6 (0.9) | 8.5 (0.8)
HbA1c ≥ 8% [Count of Participants; unit: Participants] | 106 | 51 | 157
Daily Insulin Dose [Mean (Standard Deviation); unit: units/kg] | 0.63 (0.20) | 0.59 (0.17) | 0.62 (0.19)
Previous or Current CGM Use [Count of Participants; unit: Participants] | 124 | 59 | 183
Duration of Insulin Pump Use [Mean (Standard Deviation); unit: years] | 9.5 (7.4) | 9.8 (6.8) | 9.6 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time in Range 70-180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: Comparing intervention group with control group during the 13-week study phase
Population: Subjects are included in the Primary Endpoint Analysis even if data for one period is missing.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 62
Percentage of time
  Baseline: number analyzed (Participants) | 129 | 61
  Baseline | 43.9 (14.0) | 41.3 (14.6)
  13 Weeks | 61.2 (11.2) | 43.8 (14.5)

2. Secondary Outcome: Percent of Time <54 mg/dL (Non-inferiority)
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Population: Subjects are included in the Secondary Endpoint Analysis even if data for one period is missing.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 62
Percentage of time
  Baseline: number analyzed (Participants) | 129 | 61
  Baseline | 0.32 (0.53) | 0.42 (0.91)
  13 Weeks | 0.23 (0.23) | 0.37 (0.53)

3. Secondary Outcome: Percent of Time >180 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Population: Subjects are included in the Secondary Endpoint Analysis even if data for one period is missing.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 62
Percentage of time
  Baseline: number analyzed (Participants) | 129 | 61
  Baseline | 54.4 (14.7) | 57.1 (15.5)
  13 Weeks | 37.6 (11.4) | 54.5 (15.4)

4. Secondary Outcome: Mean Glucose
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Population: Subjects are included in the Secondary Endpoint Analysis even if data for one period is missing.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 62
mg/dL
  Baseline: number analyzed (Participants) | 129 | 61
  Baseline | 200.0 (29.5) | 204.2 (30.7)
  13 Weeks | 173.7 (19.7) | 199.8 (30.3)

5. Secondary Outcome: Change in HbA1c
Description: Measures device effectiveness
Time Frame: Baseline compared to end of study visit (Day -30 to Day 90)
Population: Subjects are included in the Secondary Endpoint Analysis even if data for one period is missing.
Measure: Mean (Standard Deviation); unit: percentage of HbA1C
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 119 | 55
percentage of HbA1C | -1.24 (0.75) | -0.68 (0.93)

6. Secondary Outcome: Percent of Time <70 mg/dL
Description: Glucose metric from study continuous glucose monitoring system
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Population: Subjects are included in the Secondary Endpoint Analysis even if data for one period is missing.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 62
Percentage of time
  Baseline: number analyzed (Participants) | 129 | 61
  Baseline | 1.66 (1.79) | 1.66 (2.25)
  13 Weeks | 1.18 (0.86) | 1.75 (1.68)

7. Secondary Outcome: Change in Diabetes Distress Scale for Adults With Type 1 Diabetes (T1-DDS) Total Score
Description: A questionnaire that measures seven critical dimensions of distress (28-item scale with 6 choices that range from 1 (Not a Problem) to 6 (A Very Serious Problem)). The total score can range from 1 to 6, with a lower score indicating a better outcome.
Time Frame: Baseline compared to end of study visit (Day -14 to Day 90)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 130 | 60
score on a scale | -0.30 (0.50) | -0.20 (0.47)

8. Secondary Outcome: Change in Hypoglycemic Confidence Scale (HCS) Total Score
Description: A questionnaire that examines the degree to which people with diabetes feel able, secure, and comfortable regarding their ability to stay safe from hypoglycemic-related problems (9-item scale with 4 choices that range from 1 (Not Confident At All) to 4 (Very Confident)). The total score can range from 1 to 4, with a higher score indicating a better outcome.
Time Frame: Baseline compared to end of study visit (Day -14 to Day 90)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 60
score on a scale | 0.16 (0.52) | 0.01 (0.49)

9. Secondary Outcome: Change in Diabetes Quality of Life (DQOL)-Brief Total Score
Description: A questionnaire that assesses the relative burden of an intensive diabetes treatment regimen (15-item scale with 5 choices that range from 1 (Very Dissatisfied/All the Time) to 5 (Very Satisfied/Never)). The total score can range from 1 to 5, with a higher score indicating a better outcome.
Time Frame: Baseline compared to end of study visit (Day -14 to Day 90)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 130 | 60
score on a scale | 0.35 (0.44) | -0.02 (0.45)

10. Secondary Outcome: Proportion of Participants With T1-DDS MCID After 13 Weeks
Description: Proportion of participants achieving a minimal clinically important difference (MCID) of ≥ 0.19 points (improvement) on the T1-DDS questionnaire total score at 13 weeks compared between treatment groups
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 130 | 60
Participants | 70 | 27

11. Secondary Outcome: Proportion of Participants With DQOL-brief Clinically Meaningful Improvement After 13 Weeks
Description: Proportion of participants achieving a clinically meaningful improvement in the DQOL-brief total score after 13 weeks
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 130 | 60
Participants | 77 | 13

12. Secondary Outcome: Proportion of Participants With HCS Mean Score ≥ 3 After 13 Weeks
Description: Secondary Effectiveness Endpoint of Proportion of Participants with HCS Mean Score ≥ 3 After 13 Weeks OP5
Time Frame: Comparing intervention group with control group at the end of the 13-week study phase
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 131 | 60
Participants | 107 | 37

ADVERSE EVENTS:
Time Frame: Start time of the standard therapy (14-days prior to Study Day 1) and continued until the participant's participation ended, up to 13 weeks.
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/132 | 1/62
Other Adverse Events (participants affected / at risk) | 11/132 | 8/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=132) | Control Arm (N=62)
Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Tibia fracture requiring surgery.
Severe Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=132) | Control Arm (N=62)
Other (Investigations) | 5 (6) | 4 (4) — The 'other' events in the Omnipod 5 System group included concussion, lumbosciatica, pneumonia, shoulder pain, skin reaction and angina. The 'other' events in the Control group included laryngitis, fibula fracture, foot fracture and sciatica.
Prolonged Hyperglycemia (Endocrine disorders) | 4 (4) | 4 (5)
Hyperglycemia (Endocrine disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT05409131/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT05409131/SAP_001.pdf